CLINICAL TRIAL: NCT02291263
Title: Assessing the Immunogenicity of Intramuscular Inactivated Poliovirus Vaccine Against Type 2 With Bivalent Oral Poliovirus Vaccine in Routine Immunization
Brief Title: Immunogenicity of Intramuscular Inactivated Poliovirus Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICDDRB-RRC-PR-13097
Record Dates: First submitted 2014-11-04; First posted 2014-11-14 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Poliomyelitis
Keywords: Polio; Inactivated polio vaccine; IPV; oral polio vaccine
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): Group A will receive 3 doses of bivalent oral polio vaccine (bOPV) at 6, 10 and 14 weeks of age. Group A participants will also receive inactivated polio vaccine (IPV) at 6 weeks of age. An additional dose of IPV will be administered at 18 weeks of age.
  Interventions: Biological: bOPV/IPV (6 weeks)
- Arm B (Active Comparator): Group B will receive 3 doses of bivalent oral polio vaccine (bOPV) at 6, 10 and 14 weeks of age. Group B participants will also receive inactivated polio vaccine (IPV) at 14 weeks of age. An additional dose of IPV will be administered at 18 weeks of age.
  Interventions: Biological: bOPV/IPV (14 weeks)
- Arm C (Active Comparator): Group C will receive 3 doses of bivalent oral polio vaccine (bOPV) at 6, 10 and 14 weeks of age. Group C participants will also receive inactivated polio vaccine (IPV) at 6 and 14 weeks of age. An additional dose of IPV will be administered at 18 weeks of age.
  Interventions: Biological: bOPV/IPV (6 & 14 weeks)

INTERVENTIONS:
Biological: bOPV/IPV (6 weeks) — bOPV at 6, 10 and 14 weeks of age IPV at 6 weeks of age
  Arms: Arm A
Biological: bOPV/IPV (14 weeks) — bOPV at 6, 10 and 14 weeks of age IPV at 14 weeks of age
  Arms: Arm B
Biological: bOPV/IPV (6 & 14 weeks) — bOPV at 6, 10 and 14 weeks of age IPV at 6 and14 weeks of age
  Arms: Arm C

SUMMARY:
This study will be an open-label phase III randomized clinical trial comparing different combinations and regimens of polio vaccines. The trial will compare one and two doses of IPV administered at 6 weeks or 14 weeks or 6 and 14 weeks of age. All participants will also receive bOPV at 6, 10 and 14 weeks of age.

DETAILED DESCRIPTION:
Oral poliovirus vaccines are live attenuated viral vaccines and the vaccine virus in OPV can mutate and acquire neurovirulence causing paralysis either due to vaccine-associated paralytic polio (VAPP) or due to circulating vaccine-derived polioviruses (cVDPVs), in which the attenuated vaccine virus not only acquires the ability to cause paralysis but can also circulate similar to wild poliovirus (WPV). The potential of vaccine virus to acquire neurovirulence and cause paralytic poliomyelitis is incompatible with eradication of polio. Therefore, polio eradication will require eventual cessation of all OPVs.

The last case of WPV2 was reported in 1999 in India. Type 2 vaccine virus in tOPV is most likely to cause cVDPVs and over 80% of cVDPVs over the past decade have been cVDPV2. Of the estimated 250-500 annual VAPP cases almost 40% are due to type 2. Thus, with the eradication of WPV2 it is imperative to prioritize removal of type 2 containing OPV.

The licensing and availability of bivalent OPV (bOPV) containing type 1 and 3 offers the option of an OPV that does not contain OPV2. In April 2013, the Strategic Advisory Group of Experts on Immunization (SAGE) recommended phased cessation of OPV types starting with the switch from trivalent oral poliovirus vaccine (tOPV) to bivalent OPV (bOPV). In November 2013, SAGE recommended that countries that introduce at least one dose of IPV in the routine immunization program should administer the first dose of IPV at ≥14 weeks of age. In countries with routine immunization schedule of 6, 10 and 14 weeks of age or 2, 3 and 4 months of age, IPV would then be added to the DTP3 visit for children on schedule or administered at the first immunization visit at 14 weeks or later if children are off schedule. For countries with 2, 4 and 6 month schedule, IPV could be added either to DTP2 or DTP3 visit. SAGE also proposed that countries have the flexibility to consider alternative schedules including administering IPV earlier than 14 weeks of age or administer more than one dose of IPV.

The principal objective of pre-eradication introduction of IPV is to mitigate the risk associated with an increased susceptibility to type 2 polioviruses when bOPV is introduced. Therefore, the objective is to achieve the highest possible type 2 population immunity with IPV, which is a product of the per dose immunogenicity of IPV and the coverage achieved by IPV at that vaccination visit in routine immunization.

At present, no study has assessed immunological response against type 2 poliovirus of a single dose of IPV at 14 weeks of age, the SAGE recommended target age for IPV introduction. Furthermore, there is need to determine the immunological response with other potential alternatives for IPV introduction in routine immunization within the context of EPI schedule including immunological response with more than one dose of IPV. Also there is urgent need to document the immunogenicity of bOPV at 6, 10 and 14 weeks of age with IPV against type 1 and 3 polioviruses.

In this trial, the investigators are trying to determine the immunogenicity of alternative schedules of administering IPV other than the SAGE recommended schedule of IPV at 14 weeks of age. How does the immunogenicity of multiple doses of IPV at 6 and 14 weeks of age compare to only one dose at 14 weeks of age? How does IPV immunogenicity at 6 weeks of age compare to IPV at 14 weeks of age?

It is well established that seroconversion with multiple doses of IPV is increased by larger interval between IPV doses. A study in Cuba reported a higher type 2 seroconversion (89% vs 83%) with two doses of IPV administered 2 months apart (8 and 16 weeks of age) compared to three doses of IPV administered one month apart (6, 10 and 14 weeks of age). The proposed trial will compare 2 doses of IPV (at 6 and 14 weeks of age) to a single dose of IPV administered at either 6 or 14 weeks of age. This trial would not only assess type 2 seroconversions with IPV but also determine priming against type 2 poliovirus with the different proposed IPV schedules. Additionally, all trial participants will receive bOPV at 6, 10 and 14 weeks of age. This would permit the trial to determine type 1 and type 3 seroconversions observed with the combination of bOPV and IPV.

Setting: Study area The study will be conducted in a suburb of Dhaka in the area of Mirpur. Mirpur is one of the 14 Thanas of Dhaka city with a population of about one million in an area of 59 square kilometers. Mirpur Thana of Dhaka city is divided into 14 sections. The area is densely populated and is about 8 kilometres from icddr,b's Dhaka Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6-7 weeks of age
* Family that consents for participation in the full length of the study
* Family that is able to understand and comply with planned study procedures

Exclusion Criteria:

* Family that is unable to participate in the full length of the study
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of IPV or collection of blood by venipuncture
* Acute diarrhea, infection or illness at the time of enrollment (6-7 weeks of age) that would require infant's admission to a hospital or would contraindicate provision of OPV per country guidelines
* Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit (6 weeks of age)
* Receipt of any polio vaccine (OPV or IPV) before enrollment based upon documentation or parental recall
* Known allergy/sensitivity or reaction to polio vaccine or contents of polio vaccine
* Infants from multiple births. Infants from multiple births will be excluded to reduce the potential for contact transmission of vaccine poliovirus to siblings. The infant(s) from a multiple birth who is/are not enrolled would be likely to receive routine immunization and transmit vaccine poliovirus to the enrolled infant
* Infants from premature births (<37 weeks of gestation)

Ages: 6 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 738 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in antibody titers at 18 and 19 weeks of age compared to 6 weeks of age | Change at 18 and 19 weeks of age compared to 6 weeks of age
  The primary analytical approach will be intention-to-treat analysis. Sum of seroconversion and priming as one outcome. Seroconversion is defined as either seronegative participants (<1:8 titers) who become seropositive (≥1:8) or participants who demonstrate a 4-fold change in titers between two specimens, e.g. a change from 1:8 to 1:32 from 6 weeks to 18 weeks of age, respectively.
  Priming is defined as absence of type 2 seroconversion by 18 weeks with type 2 seroconversion at 19 weeks, i.e. seronegative participants at 18 weeks (<1:8 titers) who become seropositive at 19 weeks (≥1:8) or a 4-fold rise in type 2 antibody titers at 19 weeks compared to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Md. Khalequzzaman, MBBS, PhD, Principal Investigator — International Center for Diarrhoeal Disease Research, Bangladesh; Abhijeet Anand, MBBS, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Mirpur clinic (International Center for Diarrhoeal Disease Research, Bangladesh), Dhaka, Bangladesh